CLINICAL TRIAL: NCT03712709
Title: Prospective, Multicentre Trial to Assess the Diagnostic Accuracy of the Truenat Assays at Intended Settings of Use
Brief Title: Clinical Evaluation of the Truenat Point-of-care Tuberculosis Diagnostic Test
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Burnet Institute (Other); National Institute for Research in Tuberculosis, Chennai, India (Unknown); Universidad Peruana Cayetano Heredia (Other); Ethiopian Public Health Institute (Other Government); PD Hinduja Hospital and Medical Research Centre, Mumbai, India (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7212-03/2
Record Dates: First submitted 2018-09-27; First posted 2018-10-19 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Participant sputum may be retained for future research on TB diagnostics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Detection Group: Clinical suspicion of pulmonary TB (including cough ≥2 week and at least 1 other symptom typical of TB). Only participants who have not received any form of TB treatment within the prior 60 days will be enrolled
  Interventions: Diagnostic Test: Truenat MTB
- Drug Resistant TB Group: In addition to the criteria of the Case Detection Group, participants should also meet the following conditions: Non-converting pulmonary TB cases (category I and category II failures).
  Interventions: Diagnostic Test: Truenat MTB

INTERVENTIONS:
Diagnostic Test: Truenat MTB — The Truenat MTB (including both MTB and MTB Plus) and the MTB-RIF Dx reflex assays (Molbio Diagnostics; Bangalore, India) utilize chip-based real-time micro-PCR for detection of tuberculosis (TB) and rifampicin (RIF) resistance from DNA extracted (on a separate device) from sputum samples. The Truenat MTB assay targets a single copy gene while the MTB Plus assay combines detection of a single copy and multi-copy gene.
  Other Names: Truenat MTB Plus; Truenat MTB-RIF Dx

SUMMARY:
Consenting adults presenting with signs and symptoms compatible with pulmonary tuberculosis will be interviewed for demographic and medical information, and then will be asked to provide 3-4 expectorated sputum specimens. In the study laboratory, sputa will be tested using conventional and investigational diagnostic tests for tuberculosis and rifampin resistance.

ELIGIBILITY:
Inclusion Criteria:

Case Detection Group:

* Age 18 years or above
* Clinical suspicion of pulmonary TB (including cough ≥2 week and at least 1 other symptom typical of TB);
* Willingness to provide 3-4 sputum specimens at enrolment;
* Willingness to have a trial follow-up visit approximately 2 months after enrolment;
* Provision of informed consent.

Drug Resistant TB Group:

In addition to the criteria of the Case Detection Group, participants should also meet the following conditions:

* Non-converting pulmonary TB cases (category I and category II failures)

Exclusion Criteria:

Case Detection Group:

* Receipt of any dose of TB treatment within 60 days prior to enrolment (even if within last two days only).

Drug Resistant TB Group:

* Receipt of any dose of MDR-TB treatment within 60 days prior to enrolment (even if within last two days only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from outpatient TB clinics at district or regional health facilities. Given the important role of the private sector in India, 1 private laboratory will be included in the trial which is an MDR reference hospital.
  This is a multi-centre trial conducted in four countries: India, Peru, Papua New Guinea and Ethiopia. Countries were selected to be globally representative of the TB epidemic.
Sampling Method: Non-Probability Sample
Enrollment: 1926 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy (Sensitivity and Specificity) of the Truenat MTB assay | Day 1
  Estimate diagnostic accuracy of the Truenat assays (MTB and MTB Plus) for Mycobacterium tuberculosis (MTB) detection among individuals undergoing evaluation for pulmonary TB, using a culture reference standard

SECONDARY OUTCOMES:
Diagnostic accuracy (Sensitivity and Specificity) of the Truenat MTB-RIF Dx assay | Day 1
  Estimate diagnostic accuracy of the Truenat MTB-RIF Dx assay for RIF resistance detection among individuals undergoing evaluation for pulmonary TB and DR TB, using phenotypic/genotypic drug susceptibility testing (DST) .
Diagnostic accuracy (Sensitivity and Specificity) of the Truenat MTB assay compared to Xpert MTB/RIF | Day 1
  Compare the diagnostic accuracy of the Truenat assays (MTB and MTB Plus) to that of Xpert MTB/RIF, using a reference standard of culture for TB diagnosis and phenotypic/genotypic DST for detection of RIF resistance.
Diagnostic accuracy (Sensitivity and Specificity) of the Truenat MTB-RIF Dx assay compared to Xpert MTB/RIF | Day 1
  Compare the diagnostic accuracy of the Truenat MTB-RIF Dx assay to that of Xpert MTB/RIF, using a reference standard of culture for TB diagnosis and phenotypic/genotypic DST for detection of RIF resistance.
Time to TB detection and RIF resistance detection. | Day 1
  Assess patient important outcomes, including time to detection of TB and RIF resistance.

CONTACTS AND LOCATIONS:
Locations (4):
- EPHI, Addis Ababa, Ethiopia
- India (3):
  - State TB and Demonstration Center, Ahmedabad
  - NIRT, Chennai
  - PD Hinduja Hospital, Mumbai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nikam C, Jagannath M, Narayanan MM, Ramanabhiraman V, Kazi M, Shetty A, Rodrigues C. Rapid diagnosis of Mycobacterium tuberculosis with Truenat MTB: a near-care approach. PLoS One. 2013;8(1):e51121. doi: 10.1371/journal.pone.0051121. Epub 2013 Jan 21. PMID 23349670
- [Result] Nikam C, Kazi M, Nair C, Jaggannath M, M M, R V, Shetty A, Rodrigues C. Evaluation of the Indian TrueNAT micro RT-PCR device with GeneXpert for case detection of pulmonary tuberculosis. Int J Mycobacteriol. 2014 Sep;3(3):205-10. doi: 10.1016/j.ijmyco.2014.04.003. Epub 2014 Jun 2. PMID 26786489
- [Derived] Inbaraj LR, Daniel J, Sathya Narayanan MK, Srinivasalu VA, Bhaskar A, Scandrett K, Rajendran P, Kirubakaran R, Shewade HD, Malaisamy M, Padmapriyadarsini C, Takwoingi Y. Truenat MTB assays for pulmonary tuberculosis and rifampicin resistance in adults and adolescents. Cochrane Database Syst Rev. 2025 Mar 24;3(3):CD015543. doi: 10.1002/14651858.CD015543.pub2. PMID 40122135
- [Derived] Penn-Nicholson A, Gomathi SN, Ugarte-Gil C, Meaza A, Lavu E, Patel P, Choudhury B, Rodrigues C, Chadha S, Kazi M, Mace A, Nabeta P, Boehme C, Gangakhedkar RR, Sarin S, Tesfaye E, Gotuzzo E, du Cros P, Tripathy S, Ruhwald M, Singh M, Denkinger CM, Schumacher SG; Truenat Trial Consortium; Members of the Truenat Trial Consortium:. A prospective multicentre diagnostic accuracy study for the Truenat tuberculosis assays. Eur Respir J. 2021 Nov 4;58(5):2100526. doi: 10.1183/13993003.00526-2021. Print 2021 Oct. PMID 34049948
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229

DOCUMENTS (2):
  • Study Protocol (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03712709/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03712709/SAP_001.pdf